CLINICAL TRIAL: NCT04178850
Title: A Randomized, Double-blind, Multi-center Phase Ⅲ Comparative Study to Evaluate the Efficacy and Safety of Recombinant Human-mouse Chimeric Anti-TNF-alpha Monoclonal Antibody for Injection.
Brief Title: Clinical Comparative Study to Evaluate the Efficacy and Safety of Recombinant Anti-TNF-alpha Antibodies for Injection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GENOR GB242-002
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Folic Acid; Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GB242 (Experimental): 3mg/kg
  Interventions: Biological: GB242
- Infliximab (Active Comparator): 3mg/kg
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: GB242 — GB242: Dosing of 3 mg/kg, intravenous drip, to be completed over 120 minutes, dosing at weeks 0, 2, 6, 14 and 22, a total of 5 doses; MTX:Dosage and administration at enrollment are maintained (10~15mg/week), oral administration, a total of 30 doses; Folic acid: 5-10mg/week, oral administration, a total of 30 doses
  Other Names: MTX; Folic acid
  Arms: GB242
Biological: Infliximab — Infliximab: Dosing of 3 mg/kg, intravenous drip, to be completed over 120 minutes, dosing at weeks 0, 2, 6, 14 and 22, a total of 5 doses; MTX:Dosage and administration at enrollment are maintained (10~15mg/week), oral administration, a total of 30 doses; Folic acid: 5-10mg/week, oral administration, a total of 30 doses
  Other Names: MTX; Folic acid
  Arms: Infliximab

SUMMARY:
This study compares the similarity of the proportion of subjects who achieved ACR20 at week 30 in the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years, males or females;
2. Subjects who have confirmed rheumatoid arthritis for at least 3 months according to 2010 American College of Rheumatology Classification Criteria (amendment);
3. The active stage is met at screening: the following 3 items should be met (based on 28 joints):

   Swelling of 4 or more joints; tenderness of 6 or more joints; Tenderness of 6 or more joints; At least one of the following criteria is met: erythrocyte sedimentation rate >28mm/h or C-reactive protein >10mg/L (1mg/dl);
4. Subjects who have been treated with MTX treatment for at least 3 months before the before the use of invesetigational products and the dose remains stable (10~15mg/week) for at least 4 weeks;
5. The following DMARDs except MTX (including but not limited to chloroquine, hydroxychloroquine, gold preparation, penicillamine, sulfasalazine, azathioprine, cyclophosphamide, cyclosporin A, glucosinolate, auranofin etc.) are discontinued at least 4 weeks before the use of invesetigational products. Should any leflunomide is previously used, the subjects can be enrolled after 4 weeks after washout with cholestyramine (8g, three times per day) for 11 days. If leflunomide is discontinued 12 weeks ago, the patients can be enrolled without washout with cholestyramine.
6. If glucocorticoids are being administered before the use of invesetigational products, the dose must be stable and remains ≤10mg/d (equivalent to the dose of prednisone) for at least 4 weeks; if no glucocorticoids is used, no oral administration is given at least 4 weeks ago or no local injection is given at least 12 weeks ago.
7. The Chinese traditional patent medicine or Chinese herbal medicine for RA treatment, physical therapy, inoculation with live (attenuated) viral/ bacterial vaccines, or intravenous injection of immunoglobulin (IgG) should be discontinued at least 4 weeks before the use of the use of invesetigational products;
8. If other biological preparations are used, or the subjects participated in clinical trials of other investigational products or marketed drugs before the use of invesetigational products, an interval of at least 3 months is required.
9. Female patients of child-bearing potential have negative pregnancy test at screening; both males and females agree to adopt medically confirmed effective contraceptive measures during the entire study period and within 6 months after the end of this study.
10. Voluntarily participate in the clinical trial and sign the informed consent form;
11. Be able to understand and complete assessment forms;
12. Patients can well communicate with the investigators and complete the study as required by the study.

Exclusion Criteria:

1. The subjects received similar biological preparations (TNF inhibitors) for RA treatment within 3 months before randomization or were treated with TNF inhibitors 3 months ago, which are assessed as ineffective by the investigator.
2. Be allergic to any exicipent of the investigational products or any other murine or human-derived protein, hypersensitivity to immunoglobulin products, known to have medical history of allergic diseases or allergic constitution;
3. Body weight >100kg;
4. Subjects with rheumatoid arthritis with joint function classification of grade IV or subjects who combined to chair or bed (refer to appendix 9 for details of joint function classification);
5. Treatment with interferon within 4 weeks before the use of invesetigational products;
6. Any of the following is positive: hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), acquired immunodeficiency syndrome antibody (Anti-HIV) and anti-treponema pallidum antibody (TP-Ab);
7. Patients with known tuberculosis infection and patients with high risks for tuberculosis infection should be excluded. If patients with latent tuberculosis infection (LTBI) agree to receive preventive anti-tuberculosis therapies (appendix 5) during the study period, they can be enrolled. Or, they will be excluded.1) Known tuberculosis infection (any of the following criteria is met):

   A. Active tuberculosis infection or presence of clinical signs and symptoms of suspected tuberculosis (pulmonary or extrapulmonary);B. Presence of active tuberculosis infection involved any organ system, or symptoms of other organ systems corresponding to tuberculosis infection;C. The radiology test or other imaging tests showing evidence of previous infection at screening or within the previous 3 months (obsolete tuberculosis evidence: scars of lung and/or pleural fiber; calcification of apex of lung or other sites; pulmonary hilus and /or mediastinal lymph node lesions; decreased volume of upper lobe of lung; pulmonary cavity).2) High risks for tuberculosis infection (any of the following criteria is met): A. Known to be in close contact with active tuberculosis patients within 3 months before screening; B. Subjects with low immunologic function and with evidence showing any latent tuberculosis infection (LTBI); C. Long stay with individuals infected with tuberculosis or long stay in medical service environment or institutions with high risks for tuberculosis transmission and infection;3) If patients with latent tuberculosis infection (LTBI) agree to receive preventive anti-tuberculosis therapies (appendix 5) during the study period, they can be enrolled. Or, they will be excluded.

   LTBI is defined as no evidence showing signs or symptoms of tuberculosis infection or abnormal physical examination, and chest X-ray test (other imaging tests) results showing no evidence of tuberculosis infection, however, interferon gamma release assay (IGRA) is positive or the results of two IGRA tests are not clear;
8. Previous opportunistic infection (herpes zoster, cytomegalovirus, mycoplasma, pneumocystis carinii, histoplasma capsulatum, candida, aspergillus, mycobacterium other than mycobacterium tuberculosis etc.) within 6 months before screening;
9. Medical history of chronic infection (e.g., chronic hepatitis, chronic renal infection etc.), serious or life-threatening infection (e.g., hepatitis, pneumonitis and pyelonephritis etc.) or any current symptoms or signs indicating possible presence of infection (e.g., pyrexia, cough, urgent micturition, urodynia, abdominal pain, diarrhea, cutaneous infected wound etc.)
10. Patients who are in high risk for infection (e.g., leg ulcer, retention catheterization, persistent or recurrent chest infection and bedridden or wheelchair-bound for a long term);
11. Medical history of lymphoproliferative disorder (including lymphoma, or signs or symptoms reflecting lymphoproliferative disorders at any time); or splenomegaly;
12. Patients who previously or currently have malignant tumors within 5 years before screening (excluding adequately treated and completely cured skin basal cell carcinoma or squamous cell carcinoma, cervical in situ carcinoma);
13. Current or previous presence of congestive heart failure or medical history of congestive heart failure;
14. Current presence of interstitial lung disease or medical history of previous interstitial lung disease;
15. Current or previous presence of multiple sclerosis or other demyelinating diseases of the central nervous system or corresponding medical history of these diseases;
16. There is evidence showing that the patients have serious, progressive and uncontrolled cardiovascular, renal, hepatic, hemopoietic, gastrointestinal, endocrine, pulmonary, nervous system disorders; and other conditions who are considered unsuitable for participating in this study at the discretion of the investigator;
17. The following abnormal laboratory variables should be excluded: white blood cells (WBC) <3.0×109/L, neutrophil count (ANC)<1.5×109/L, platelet count (PLT) <100×109/L, hemoglobin (HGB) <85g/L, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the upper limit of normal (ULN), alkaline phosphatase (ALP)> 2 times the upper limit of normal (ULN), serum creatinine (Cr) > 1.5 times ULN;
18. Current or previous presence of other systemic immune diseases (e.g., systemic lupus erythematosus etc.), or inflammatory joint disease other than rheumatoid arthritis (e.g., gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy and Lyme disease etc.); Patients with rheumatoid arthritis complicated with secondary Sjogren syndrome which will not affect drug evaluation at the discretion of the investigator are allowed to be enrolled.
19. Subjects with medical history of prosthetic joint infection and the artificial joints are still in the body;
20. Subjects who received arthroplasty for more than 3 times;
21. Subjects who received organ transplantation within 6 months before screening;
22. Lactating women;
23. Subjects who have medical history of long-term alcohol abuse or drug abuse;
24. Subjects who have insufficient communication, understanding and cooperation, or subjects who have low education level, cannot understand and correctly complete corresponding forms, subjects who have history of noncompliance with doctor's instructions to receive administration, or subjects who have other conditions which may interfere with protocol compliance of subjects (e.g., subjects who have psychiatric disorders or usually travel, and lack of motivation to participate in the study);
25. Subjects who have other diseases (e.g., clinically significant symptoms or abnormal laboratory variables) which are considered unsuitable for participating in this clinical study at the discretion of the investigator; This study allows repeated screening at screening. The most recent test results prior to the first dose of all items are regarded as the baseline values.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 568 (Estimated)
Dates: Start 2017-10-13 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with ACR20 | Up to 30 weeks.
  Number of Participants with ACR20

SECONDARY OUTCOMES:
Number of Participants with ACR50 | Up to 30 weeks.
  Number of Participants with ACR50
Number of Participants with ACR70 | Up to 30 weeks.
  Number of Participants with ACR70
Number of Participants with DAS28 | Up to 30 weeks.
  Number of Participants with DAS28
Anti-Drug Antibody, ADA | Up to 30 weeks.
  Anti-Drug Antibody, ADA
AUC τ | Up to 30 weeks.
  AUC τ
C min,ss | Up to 30 weeks.
  C min,ss
C max,ss | Up to 30 weeks.
  C max,ss
C av,ss | Up to 30 weeks.
  C av,ss
T 1/2 | Up to 30 weeks.
  T 1/2
CL ss /F | Up to 30 weeks.
  CL ss /F
Adverse Effect, AE | Up to 30 weeks.
  Adverse Effect, AE
Serious Adverse Efect, SAE | Up to 30 weeks.
  Serious Adverse Efect, SAE

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Ph.D, Principal Investigator — Peking University People Hospital
Locations (1):
- Peking University People Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No